CLINICAL TRIAL: NCT04201821
Title: Fecal Microbial Transplantation (FMT) For the Treatment of Fecal Incontinence in Women
Brief Title: Fecal Microbial Transplantation for the Treatment of Fecal Incontinence in Women
Acronym: FMT for FI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 834196
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMT Administration (Experimental): This is a single arm study in which all eligible participants will receive FMT.
  Interventions: Biological: fecal microbial transplantation (FMT)

INTERVENTIONS:
Biological: fecal microbial transplantation (FMT) — Fecal microbial transplantation (FMT) is the infusion of intestinal microbiota from healthy donors.

SUMMARY:
Open label pilot study assessing FMT to treat fecal incontinence in women 50 years of age and older.

DETAILED DESCRIPTION:
Fecal incontinence, also known as accidental bowel leakage, is a common condition that is an immense burden to older women, caregivers, and the health care system. The overall goal of this study is to gather pilot data in order to conduct a future randomized controlled trial (RCT) for a novel treatment for fecal incontinence in older women utilizing fecal microbial transplantation (FMT). The investigator's hypothesis is that infusion of intestinal microbiota from healthy donors to older women with fecal incontinence will increase microbial diversity, reduce symptom severity, and improve quality of life. This study is a single arm, open-label clinical trial of FMT for the treatment of fecal incontinence refractory to conservative management. The investigators will measure the impact of FMT on change in symptom severity and quality of life and stool microbial diversity at 4 and 12 weeks after FMT.

ELIGIBILITY:
Inclusion Criteria:

* Women 50 years of age and older with self-reported fecal incontinence defined as:
* Uncontrolled bothersome loss of liquid or solid fecal material that occurs at least weekly over the last 3 months and
* Failure of response to conservative management using fiber, diet modification, supervised pelvic floor exercises
* Baseline St. Mark's score of greater than or equal to 12
* Intolerance, unwillingness or inadequate response to constipating medications
* Self-reported current negative colon cancer screening based on the 2016 US preventive Services Task Force recommendation (applies to participants age 50-75). N/A if participant is over 75
* Able and willing to sign the informed consent form and agree with study procedures

Exclusion Criteria:

* Known food allergy that could lead to anaphylaxis
* Contraindications to naso-gastric tube placement including:
* Recent mid-face trauma
* History basilar skull fracture
* Recent ENT surgery
* Known coagulation abnormalities
* Esophageal varices and/or esophageal strictures
* Untreated prolapse beyond the hymen
* History of Inflammatory Bowel Disease (does not include IBS)
* Unrepaired rectovaginal fistula/chronic 4th degree laceration
* Full thickness rectal prolapse
* History of congenital anorectal malformation
* History of bowel resection surgery for any indication
* Minor anal procedures within 6 months for treatment of accidental bowel leakage (ABL) (injection of bulking agent or radiofrequency energy) or ligation of hemorrhoids
* Prior pelvic or abdominal radiation
* Diagnosis of cancer of the descending colon or anus

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uduak U Andy, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 Subjects were enrolled. 2 subjects dropped out prior to administration of the investigational product. 8 subjects were treated with the investigational product.
Groups:
- FMT Administration: This is a single arm study in which all eligible participants will receive FMT.
  Fecal microbial transplantation (FMT) is the infusion of intestinal microbiota from healthy donors.
Period: Overall Study
Arm/Group | FMT Administration
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | FMT Administration
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Show Significant Improvement at 4 Weeks After FMT, and Will be Maintained at 12 Weeks, Relative to Baseline Using the St. Mark's Vaizey Score, a Measure of Fecal Incontinence Severity.
Description: The St Marsk's Viazy score is a validated patient-reported instrument used to measure fecal incontinence severity. Score ranges from 0-24 with a decrease in the score representing an improvement. A subject has clinical improvement if they have demonstrated a sustained decrease of 4-5 points between the 4-week and 12-week measurements.
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Administration
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Count of Participants With Adverse Events.
Description: Frequency of adverse events, serious adverse events, and adverse events of special interest (including allergic reaction and gastrointestinal symptoms).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Administration
Number analyzed (Participants) | 8
Participants | 6

3. Secondary Outcome: Number of Subjects That Have an Improved Quality of Life at 4 and 12 Weeks, Measured by the FIQL Scale.
Description: The FIQL is a valid and reliable 29-item questionnaire designed to evaluate the impact of FI on four aspects (domains) of patients' quality of life: lifestyle; coping behavior; depression or self-perception; and level of embarrassment. Domain scores range from 1-4 (higher scores indicating better quality of life). An improvement in the score of 1 (one) within each domain would indicate an improvement in the quality of life.
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Administration
Number analyzed (Participants) | 8
Participants | 0

4. Secondary Outcome: Count of Participants That Demonstrate Microbial Engraftment Following Fecal Microbial Transplantation and Demonstrate Clinical Improvement.
Description: Concentration of Microbiota present at baseline vs at week 4 in subjects that demonstrate a significant improvement at 4 weeks after FMT, relative to baseline using the St. Mark's Vaizey score.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Administration
Number analyzed (Participants) | 8
Participants | 0

5. Other Pre Specified Outcome: Count of Participants That Demonstrate Engraftment Following Fecal Microbial Transplantation.
Description: Concentration of microbiota at baseline vs concentration of microbiota at 4 weeks.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Administration
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Frequency of adverse events, serious adverse events, and adverse events of special interest (including allergic reactions and gastrointestinal symptoms)
Arm/Group | FMT Administration
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT Administration (N=8)
Abdominal Bloating (Gastrointestinal disorders) | 1 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Belching (Gastrointestinal disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 4 (10)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4)
Rectal Hemorrhage (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
General Disorder and administrative site conditions - Other - nasal irritation (General disorders) | 1 (1)
General disorders and administration site conditions - Other - nostril pain (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT04201821/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT04201821/ICF_001.pdf